CLINICAL TRIAL: NCT01245283
Title: Comparative Resistance Exercise Effect on Knee Osteoarthritis Pain, Functional Impairment and Cartilage Turnover
Brief Title: Resistance Exercise and Knee Osteoarthritis Pain, Functional Impairment and Cartilage Turnover
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 614-2009
Record Dates: First submitted 2010-11-05; First posted 2010-11-22 (Estimated); Results first posted 2014-10-08 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-11

CONDITIONS: Knee Osteoarthritis
Keywords: knee; osteoarthritis; pain; function; impairment
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Wait-list Non-exercise Control (CON) (Active Comparator): Subjects will continue to participate in their normal activities and clinical care during the four month study period if assigned to this group.
  Interventions: Other: normal activities and clinical care
- Concentric Focused RX (CRX) (Active Comparator): Training protocol for 1 set of each exercise will be completed - leg press, leg curl, leg extension, chest press, seated row, overhead press, triceps dip, biceps curl, and calf press.
  Interventions: Other: Concentric Focused Resistance Exercise
- Eccentric Focused RX (ERX) (Active Comparator): The Human Dynamics Laboratory features prototype equipment that increases resistance loads during the eccentric phase of the contraction while "assistance" is provided by the machine during the concentric phase. One set of each exercise - leg press, leg curl, leg extension, chest press, seated row, overhead press, triceps dip, biceps curl, and calf press.
  Interventions: Other: Eccentric Focused Resistance Exercise

INTERVENTIONS:
Other: normal activities and clinical care — Subjects will continue to participate in their normal activities and clinical care during the four month study. Telephone contact will be made weekly to encourage adherence to the knee management guidelines
  Arms: Wait-list Non-exercise Control (CON)
Other: Concentric Focused Resistance Exercise — Two resistance exercise sessions per week; 1 set of 10-12 repetitions of each exercise will be completed - leg press, leg curl, leg extension, chest press, seated row, overhead press, triceps dip, biceps curl, and calf press.
  Arms: Concentric Focused RX (CRX)
Other: Eccentric Focused Resistance Exercise — Two resistance exercise sessions per week; 1 set of 10-12 repetitions of each exercise will be completed - leg press, leg curl, leg extension, chest press, seated row, overhead press, triceps dip, biceps curl, and calf press.
  Arms: Eccentric Focused RX (ERX)

SUMMARY:
The purpose of this study is to determine if a 4 month resistance exercise program can reduce knee osteoarthritis pain functional impairment and cartilage turnover.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis (OA) of the knee for >6 months
* moderate to severe pain immediately following a 50-foot walk
* knee pain primarily due to tibiofemoral OA and not from patellofemoral OA
* bilateral standing anterior-posterior radiograph demonstrating grade 2 or 3 OA of the target knee
* willing and able to participate in regular exercise for four months
* free from musculoskeletal limitations that would preclude resistance exercise participation
* free of abnormal cardiovascular responses during the screening graded maximal walk test

Exclusion Criteria:

* unable to walk
* regular resistance exercise training (>3X week) within the past 6 months
* specific low back pain or acute back injury
* spinal stenosis that precludes walking one block due to neurogenic claudication
* any major injury to either knee within the prior 12 months
* any surgery to either knee within the last 12 months
* lumbar radiculopathy
* vascular claudication
* significant anterior knee pain due to diagnosed isolated patella-femoral syndrome or chondromalacia in either knee
* have had corticosteroid or viscosupplement injections within three months of study participation
* have added new over the counter or prescription pain medication within two months of study participation

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin R Vincent, M.D. Ph.D., Principal Investigator — University of Florida Department of Orthopaedics and Rehabilitaion
Locations (1):
- UF&Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wait-list Non-exercise Control (CON) | Concentric Focused RX (CRX) | Eccentric Focused RX (ERX)
Started | 32 | 28 | 30
Completed | 18 | 17 | 19
Not Completed | 14 | 11 | 11
Not completed — Lost to Follow-up | 14 | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wait-list Non-exercise Control (CON) | Concentric Focused RX (CRX) | Eccentric Focused RX (ERX) | Total
Number analyzed (Participants) | 32 | 28 | 30 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (7.1) | 69.5 (6.5) | 66.8 (5.4) | 68.27 (6.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 21 | 62
  Male | 10 | 9 | 9 | 28
Region of Enrollment [Number; unit: participants]
  United States | 32 | 28 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC Score); Change From Baseline at 4 Months
Description: The WOMAC is a standard, multidimensional, self-administered functional-health status instrument for patients with lower limb OA. Subjects will complete the self-assessment at the time intervals indicated to document any change in their perception of their functional health status.
  Scale for Total score: the higher score means the worst the function and pain Total WOMAC scores will have a range of 0 to 96 (best and worst scores possible).
  0-20 Womac pain (0= best, 20=worst) 0-8 Womac stiffness (0= best, 8=worst) 0-68 Womac functional (0= best, 68=worst) 0-96 Womac Total (0= best, 96=worst)
Time Frame: Baseline, 4 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wait-list Non-exercise Control (CON) | Concentric Focused RX (CRX) | Eccentric Focused RX (ERX)
Number analyzed (Participants) | 32 | 28 | 30
units on a scale
  WOMAC total baseline | 27.1 (12.6) | 33.3 (14.1) | 28.9 (11.6)
  WOMAC total 4 months | 26.7 (20) | 23 (13.7) | 19.9 (14.0)
  WOMAC Knee pain baseline | 4.3 (2.2) | 5.4 (2.9) | 6.1 (2.7)
  WOMAC Knee pain 4 months | 4.1 (3.0) | 3.9 (3.3) | 3.4 (3.0)
  WOMAC Knee stiffness baseline | 3.8 (1.8) | 4.1 (1.5) | 3.5 (1.6)
  WOMAC Knee stiffness 4 months | 3.7 (2.1) | 3.1 (1.6) | 3.1 (2.2)
  WOMAC Knee physical function baseline | 18.9 (9.8) | 24.4 (11.1) | 19.2 (8.4)
  WOMAC Knee physical function 4 months | 18.7 (16.3) | 15.9 (9.6) | 13.3 (9.6)

2. Secondary Outcome: Six Minute Walk Test; Change From Baseline at 4 Months
Description: Each participant will walk at a self-selected pace in the lab around a pre-measured loop for a period of six minutes. Subjects will complete the walk test at the time intervals indicated to document any change. 6 minute walk test is a baseline and 4 month post intervention measurement. It is used to measure distance covered while walking during 6 minutes.
Time Frame: Baseline, 4 Months
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Wait-list Non-exercise Control (CON) | Concentric Focused RX (CRX) | Eccentric Focused RX (ERX)
Number analyzed (Participants) | 32 | 28 | 30
feet
  Six Minute Walk Baseline | 1556 (342) | 3600 (1181) | 4652 (1520)
  Six Minute Walk 4 months | 1640 (370) | 3496 (1308) | 4643 (1127)

3. Secondary Outcome: Chair Rise Time and Stair Climb Time; Change From Baseline at 4 Months
Description: Functional abilities related to moving body weight will be captured using two standard tests, the chair rise time and stair climb time. Subjects will complete the tests at the time intervals indicated to document any change in their functional abilities.
Time Frame: Baseline, 4 Months
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Wait-list Non-exercise Control (CON) | Concentric Focused RX (CRX) | Eccentric Focused RX (ERX)
Number analyzed (Participants) | 32 | 28 | 30
Seconds
  Chair Rise Time baseline | 1.5 (1.1) | 1.2 (0.7) | 1.2 (0.6)
  Chair Rise Time 4 months | 0.7 (0.3) | 0.8 (0.3) | 1.6 (3.8)
  Stair Climb Time baseline | 6.2 (2.9) | 5.3 (3.1) | 4.3 (1.5)
  Stair Climb Time 4 months | 7.3 (3.5) | 5.3 (1.8) | 5.1 (1.8)

4. Secondary Outcome: Leg Press Test; Change From Baseline at 4 Months
Description: Each participant will do a one repetition maximum. Participants will perform a leg press. The leg press is a weight training exercise in which the individual pushes a weight or resistance away from them using their legs.
Time Frame: Baseline, 4 Months
Measure: Mean (Standard Deviation); unit: foot x pounds
Arm/Group | Wait-list Non-exercise Control (CON) | Concentric Focused RX (CRX) | Eccentric Focused RX (ERX)
Number analyzed (Participants) | 32 | 28 | 30
foot x pounds
  Leg Press Baseline | 319 (116) | 374 (99) | 327 (116)
  Leg Press 4 months | 399 (109) | 357 (115) | 412 (97)

5. Secondary Outcome: Leg Extensions Test; Change From Baseline at 4 Months
Description: Each participant perform a one repetition maximum . Participants will perform a leg extension which is a resistance weight training exercise that targets the quadriceps muscle in the legs. The exercise is done using a machine called the Leg Extension Machine. This resistence is measured in pounds.
Time Frame: Baseline, 4 Months
Measure: Mean (Standard Deviation); unit: foot x pounds
Arm/Group | Wait-list Non-exercise Control (CON) | Concentric Focused RX (CRX) | Eccentric Focused RX (ERX)
Number analyzed (Participants) | 32 | 28 | 30
foot x pounds
  Leg Extention Baseline | 147 (58) | 186 (97) | 174 (104)
  Leg Extention 4 months | 181 (87) | 167 (91) | 191 (89)

6. Secondary Outcome: Leg Curl Test; Change From Baseline at 4 Months
Description: Each participant will perform a one repetition maximum. Participant will perform a leg curl which is an isolation exercise that targets the hamstring muscles. The exercise involves flexing the lower leg against resistance towards the buttocks. This resistence is measured in pounds.
Time Frame: Baseline, 4 Months
Measure: Mean (Standard Deviation); unit: foot x pounds
Arm/Group | Wait-list Non-exercise Control (CON) | Concentric Focused RX (CRX) | Eccentric Focused RX (ERX)
Number analyzed (Participants) | 32 | 28 | 30
foot x pounds
  Leg Curl Baseline | 154 (42) | 168 (57) | 155 (63)
  Leg Curl 4 months | 182 (63) | 166 (53) | 175 (49)

7. Secondary Outcome: Chest Press; Change From Baseline at 4 Months
Description: Each participant will perform a one repetition maximum. Participants will perform a chest press which is an upper body strength training exercise that consists of pressing a weight upwards from a supine position. This resistence is measured in pounds.
Time Frame: Baseline, 4 Months
Measure: Mean (Standard Deviation); unit: foot x pounds
Arm/Group | Wait-list Non-exercise Control (CON) | Concentric Focused RX (CRX) | Eccentric Focused RX (ERX)
Number analyzed (Participants) | 32 | 28 | 30
foot x pounds
  Chest Press Baseline | 170 (70) | 184 (137) | 167 (103)
  Chest Press 4 months | 199 (117) | 170 (117) | 174 (123)

8. Secondary Outcome: Shoulder Press Test; Change From Baseline at 4 Months
Description: Each participant will perform a one repetition maximum. Participants will perform the shoulder press which is a weight training exercise, typically performed while standing, in which a weight is pressed straight upwards from the shoulders until the arms are locked out overhead. This resistence is measured in pounds.
Time Frame: Baseline, 4 Months
Measure: Mean (Standard Deviation); unit: foot x pounds
Arm/Group | Wait-list Non-exercise Control (CON) | Concentric Focused RX (CRX) | Eccentric Focused RX (ERX)
Number analyzed (Participants) | 32 | 28 | 30
foot x pounds
  Shoulder Press Baseline | 158 (56) | 158 (96) | 152 (86)
  Shoulder Press 4 months | 190 (92) | 153 (87) | 147 (90)

9. Secondary Outcome: Seated Row Test; Change From Baseline at 4 Months
Description: Each participant will perform a one repetition maximum. Participants will do a seated row test which is pulling on a cable to lift weight from a seated row position. This resistence is measured in pounds.
Time Frame: Baseline, 4 Months
Measure: Mean (Standard Deviation); unit: foot x pounds
Arm/Group | Wait-list Non-exercise Control (CON) | Concentric Focused RX (CRX) | Eccentric Focused RX (ERX)
Number analyzed (Participants) | 32 | 28 | 30
foot x pounds
  Seated Row Baseline | 195 (64) | 194 (88) | 175 (79)
  Seated Row 4 months | 215 (99) | 219 (88) | 193 (107)

ADVERSE EVENTS:
Arm/Group | Wait-list Non-exercise Control (CON) | Concentric Focused RX (CRX) | Eccentric Focused RX (ERX)
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/28 | 1/30
Other Adverse Events (participants affected / at risk) | 2/32 | 2/28 | 1/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wait-list Non-exercise Control (CON) (N=32) | Concentric Focused RX (CRX) (N=28) | Eccentric Focused RX (ERX) (N=30)
Broken hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Wait-list Non-exercise Control (CON) (N=32) | Concentric Focused RX (CRX) (N=28) | Eccentric Focused RX (ERX) (N=30)
Subject inability to complete the maximum exercise test (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 — Not related to study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No